CLINICAL TRIAL: NCT04344353
Title: Analysis and Comparative Evaluation of Aortic Calcium by Computed Tomography and Histopathology in Patients With Aortic Stenosis
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Maria Elena Soto, MsC and PhD, Deputy of the Immunology Department., Instituto Nacional de Cardiologia Ignacio Chavez
Other Study IDs: 19-1139
Record Dates: First submitted 2020-04-04; First posted 2020-04-14 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Aortic Calcification Valve; Aortic Valve Stenosis
Keywords: Aortic valve stenosis; Computed Tomography; Histopathology analysis
MeSH Terms: conditions — Aortic Valve, Calcification of; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A 5-micron segment of the aortic valve, obtained by cardiothoracic surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates and compares aortic calcium by computed tomography and histopathology in patients with aortic stenosis.

DETAILED DESCRIPTION:
1. Title

   Analysis and comparative evaluation of aortic calcium by computed tomography and histopathology in patients with aortic stenosis.
2. Background.

   Calcified aortic valve disease (CAVD) was initially considered to be a passive degeneration of the extracellular matrix (EM). Recent studies have shown that within the development of the damage mechanism there is complexity and it is an active (1) and degenerative process where genetic, environmental and epigenetic phases overlap and interact leading to hemodynamic changes in blood flow, endothelial dysfunction and metabolic disorders that lead to low-density lipoprotein cholesterol deposits in the ME where at the same time there is an underlying infiltration of macrophages, oxidative stress, and release of pro-inflammatory cytokines. (2) However, although there are several theories of damage, and some of them are attributed to a diversity of origin such as genetic, congenital, infectious, and degenerative. Finally, the dynamic and functional impact of the heart affects equally. It leads to organic deterioration when the AD reaches clinical and echocardiographic criteria of severity, and the only therapeutic option is the change or replacement of the aortic valve.

   The participation of imaging methods such as computerized tomography about to the concerning the aortic valve through the measurement of the aortic calcium score (AVC-CT) as a method to determine the severity of aortic stenosis (AS) in those cases where echocardiographic measurements are conflicting, allows us to see the interest in defining this problem through different angles of investigation (7). In AD, progressive calcification is the trigger factor that also predominantly leads to aortic valve obstruction. (3) Currently, such calcification can be easily quantified using the same acquisition protocol and Agatston Scoring Method as used for a coronary artery calcium scan and is particularly attractive because it provides an assessment of the severity of AD, which is independent of the geometry and ventricular ejection fraction. Advances in the field of CT CVA measurement have been demonstrated in the last decade and are closely associated with hemodynamic measurements of moderate to severe AD in Doppler echocardiography, however, until recently, significant over-positioning of calcium from the aortic valve area among patients with hemodynamically severe AD and those with non-severe AD made it challenging to implement in clinical practice.

   This development has generated significant interest in the use of CT-CVA as an alternative and complementary assessment of the severity of AD, especially in patients with discordant echocardiographic findings. (11) In fact: 1) CVA is strongly but non-linearly associated with hemodynamic measures of severity in moderate to severe AD (12). Thus, the determination of CVA may help discriminate severe AD from non-severe AD in patients with discordant findings measured by echocardiography, and 3) in patients with moderate to severe AD, CVA is also likely associated with faster progression of AD and with survival. However, it should be mentioned that the analysis of that series did not make adjustments to the calcium measured in the patients' coronary artery. Although the CVA score has been recommended in the European Society of Cardiology Guidelines to confirm the severity of AD in the following conditions 1) patients with low left ventricular ejection fraction (LVEF), gradient and low flow, in which dobutamine stress echocardiography is inconclusive and 2) patients with low gradient AD and preserved LVEF, and this is not yet part of the American Heart Association (AHA) and American College of Cardiology (ACC) guidelines (13).

   So it has been suggested that clinical applicability should be established, so what are the next steps? While the reproducibility of coronary calcium quantification by multidetector CT has been tested for various workstation platforms before, (14,15) the same has not been done so far for CVA quantification through variability with standard Gold through the histopathological study and determine the variability of the CVA score measured by CT by determining its relationship through the flow and gradient status of patients with AD and define what implications can be suggested for the patient's treatment(13,16)
3. Problem statement.

   There is a high prevalence of aortic valve calcification in patients who are subjected to valve change regardless of the cause (genetic, congenital, or degenerative structural malformation). Early identification of calcification in these patients is critical since they will receive a valve change that is likely to return to dysfunction if there is no history of the type of damage with or without preceding valve calcification. Currently, there is controversy about the ideal time to initiate valve therapy, as it has not been possible to identify those patients who will develop significant valve calcification. However, little is known about the relationship between the new imaging methods that are promising for measuring it and its correlation with standard gold, that is, what is quantified at the histopathological level.

   3.1. Justification.

   Magnitude: The global prevalence of aortic stenosis is 0.3-0.5% and 2-7% in >65 years and of valvular calcification. According to its definition and criteria to classify valve stenosis, up to 30% will require aortic valve change due to valve insufficiency.

   Significance: In the last two decades, the incidence of aortic valve insufficiency has increased exponentially and has been associated with unfavorable outcomes.

   Vulnerability: Currently, the cornerstone of aortic stenosis management includes prevention and early support management. The identification of calcification has not been entirely clear either through laboratory parameters or about to with concerning risk factors, which are inadequate and late. Early detection and intervention of calcification during the disease can improve the prognosis if it is recognized early.

   Feasibility: The study will be carried out in the two departments of Immunology through Dr. Soto who will coordinate the research) (Cardiovascular Medicine through Dr. Israel Pérez Torres who will evaluate calcification and histological changes in the valve tissue) (Pathology through Dr. Aranda who will manage and treat the valve samples) and the Image Department coordinated by Dr. Sergio Críales Vera who will quantify the valve calcium). All departments are recognized for their extensive participation in research.

   The study of the pathogenesis of persistent inflammatory damage in aortic stenosis in relation to the type of prosthesis will lead in the future to evaluate if it is a factor involved in the recurrent damage in stenosis, calcification, and deterioration. In the last decades in Mexico, the demographic transition increased the number of people over 65 years old, the population in which the most significant complication of valve dysfunction has been seen. However, regardless of age and etiology, this is currently a population group with significant expansion and is expected to triple by 2030. This inflammatory damage will increase the prevalence of aortic stenosis, and therefore more patients will require valve replacement surgery.

   Our Institute is a national reference hospital that attends a significant number of patients with aortic stenosis, among others. Of the valves that are implanted, a quarter is manufactured at the Institute. Therefore, evaluating processes highly related to valve dysfunction such as calcification is a priority and is considered a health problem that requires prevention.

   3.2. Research question.

   In patients who have undergone aortic valve surgery, will the quantification of calcium using the 4D computerized tomography method have a reasonable correlation with that measured by histopathology, and will it also allow it to be proposed as an early predictor of dysfunction?
4. Hypothesis.

   Working hypothesis (H1): The quantifiable assessment of valve calcium by CT is similar to that measured by histopathology and predicts early valve dysfunction.

   Null hypothesis (H0): The quantifiable assessment of calcium by CT scan is different from that measured by histopathology and does not predict early valve dysfunction.
5. Methodology.

   5.1. Study design.

   Cohort, observational, comparative, and prospective study.

   5.2.5. Elimination criteria.

   a) Not having an adequate sample or staining of the valve tissue.

   5.3. Sample size.

   For the calculation of the sample size, a determination of the sample size (two tails) shall be made, taking into account the means and standard deviation (SD) of the items corresponding to each one. All patients who meet the inclusion criteria described above shall be considered for evaluation during the period 2017-2020.

   5.4. Data collection technique

   Data collection will be divided into three stages:

   Pre-surgical:

   Once the study population has been identified, a personal interview will be conducted, the objective of the study will be explained to the patient, and informed consent will be obtained. Various echocardiographic parameters will be collected for each patient (pre-surgical echocardiogram). The study of the valve, which is requested before surgery, will be analyzed in a tomography scan, and this is the one that will be used to measure the calcium.

   Post-surgery

   Employing the sample of the valve tissue obtained from the surgery, the appropriate cuts and stains for the measurement of the calcium will be requested.

   Echocardiographic study.

   The echocardiographic study performed will be re-evaluated by two expert echocardiographers following current recommendations.16 The Philips iE33 xMATRIX (Philips, Andover Massachusetts) ultrasound system with X5-1 transducer. The dimensions of the left ventricle will be quantified in the long parasternal axis; the volumes of the left atrium and left ventricle will be calculated with the Simpson method. The aortic valve area will be estimated with the continuity equation. The mass of the LV was estimated with the Devereaux method.17 The mean and maximum transvalvular aortic gradients will be acquired in the apical projection of three or five chambers, where a suitable continuous Doppler spectrum and the highest transaortic velocity were obtained. The pulmonary artery systolic pressure will be estimated by adding the right atrial pressure to the tricuspid insufficiency gradient.

   Computed tomography evaluation.

   The study was performed with a multidetector with double energy source of 256 cuts definition Flash Medical Systems Forcheim Germany (128 x 2), performing prospective additive in the best diastolic phase (65-70 %), with 3 mm thick reconstructions and 3mm spacing with Kernel B 35f filter and visual field adjusted only to the heart. The images were processed on a workstation (SmartScore by Syngo via, Waukeesha WI Electronics for Medicine. The results were expressed in Agatston units. The study was carried out without a contrast medium and with a radiation equivalent to 1.0 mSv.

   Tissue evaluation

   Histological technique.

   A 5-micron segment of the aortic valve, obtained by cardiothoracic surgery, was washed in 0.9% NaCl for 30 seconds immediately after the tissues were fixed by immersion in phosphate buffer with 10% formalin (pH 7.4) for 24 hours. Histological sections of the aortic valve were processed according to conventional histological procedures using Von Kossa staining. The technique is based on the reaction of silver nitrate in the presence of a reducing agent, usually, hydroquinone, resulting in insoluble silver phosphate that can be seen under the microscope in black. Histological sections were analyzed using a Carl Zeiss light microscope (Carl Zeiss, West Germany, Germany) (model 63,300) equipped with a Tucsen digital camera (9 megapixels) with TSview 7.1 software (Tucsen Imaging Technology Co., Ltd. Chuo, Japan, at 25x magnification. The photomicrographs were analyzed by densitometry using Sigma Scan Pro 5 Systat Software Inc. San Jose, California, CA, USA. Density values are expressed as pixel units.
6. Statistical analysis plan.

Categorical variables were expressed as proportions, continuous variables as means with standard deviation or median with interquartile range according to the distribution. Comparisons will be made for categorical variables with Chi-square or Fisher exact test and dimensional variables with Student t or Mann-Whitney U. Correlations with Pearson's r for quantitative variables or Spearman's rho for qualitative variables. Related samples were analyzed with ANOVA for repeated measurements and Friedman's test according to distribution with post-hoc analysis to identify differences between groups. The diagnostic test study will include the ROC curve to analyze cut-off points. The p-value of statistical significance was established to be less than 0.05 at two-tailed. Statistical analysis was performed with SPSS version 22 software (SPSS Inc. Chicago, Illinois).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are candidates for aortic valve replacement.
2. Age greater than or equal to 18 years of age.
3. Both genders.
4. With any associated comorbidity
5. Any etiology
6. Hospitalized and with an echocardiographic study showing the variables to be studied
7. Informed Consent.

Exclusion Criteria:

1. Patients who have previously undergone other aortic valve surgery
2. Patients who have received contrast medium ≤24 hours.
3. Patients on hemodialysis.
4. Patients with infection.
5. Patients with cancer.
6. Patients with autoimmune diseases.
7. Pregnant women.
8. Patients who refuse to be included.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population will be the patients of the Instituto Nacional de Cardiología "Ignacio Chávez." The eligible population shall consist of patients from that Institute who have been diagnosed with severe aortic stenosis and who are in the hospitalization sectors and where aortic valve replacement with a mechanical or biological prosthesis is planned. Sampling: With a non-probabilistic sequential (consecutive) technique.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
The quantifiable assessment and comparison of aortic valve calcium. | 2 days
  The study of the valve, which is requested before surgery, will be analyzed in a tomography scan. The study will be performed with a multidetector with a double energy source of 256 cuts definition Flash Medical Systems Forcheim Germany (128 x 2). The images were processed on a workstation (SmartScore by Syngo via, Waukeesha WI Electronics for Medicine). The results were expressed in Agatston units. The study was carried out without a contrast medium and with a radiation equivalent to 1.0 mSv.
  Employing the sample of the valve tissue obtained from the surgery, a 5-micron segment of the aortic valve, was washed in 0.9% NaCl for 30 seconds immediately after the tissues were fixed by immersion in phosphate buffer with 10% formalin (pH 7.4) for 24 hours. The histopathological sample will be assessed by the head of the pathology department, which will result in the percentage of calcium observed.

SECONDARY OUTCOMES:
The quantifiable assessmen and comparisont of valve calcium with photomicrographs. | 7 days
  Histological sections were analyzed using a Carl Zeiss light microscope (Carl Zeiss, West Germany, Germany) (model 63,300) equipped with a Tucsen digital camera (9 megapixels) with TSview 7.1 software (Tucsen Imaging Technology Co., Ltd. Chuo, Japan, at 25x magnification. The photomicrographs were analyzed by densitometry using Sigma Scan Pro 5 Systat Software Inc. San Jose, California, CA, USA. Density values are expressed as pixel units.
  The pixel values obtained will be compared with the calcium score obtained by computed tomography and the result provided by the pathologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional Ignacio Chavez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access will be reviewed by an external independent review panel. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Background] Otto CM, Kuusisto J, Reichenbach DD, Gown AM, O'Brien KD. Characterization of the early lesion of 'degenerative' valvular aortic stenosis. Histological and immunohistochemical studies. Circulation. 1994 Aug;90(2):844-53. doi: 10.1161/01.cir.90.2.844. PMID 7519131
- [Background] Soto ME, Salas JL, Vargas-Barron J, Marquez R, Rodriguez-Hernandez A, Bojalil-Parra R, Perez-Torres I, Guarner-Lans V. Pre- and post-surgical evaluation of the inflammatory response in patients with aortic stenosis treated with different types of prosthesis. BMC Cardiovasc Disord. 2017 Apr 14;17(1):100. doi: 10.1186/s12872-017-0526-1. PMID 28410571
- [Background] Pawade TA, Newby DE, Dweck MR. Calcification in Aortic Stenosis: The Skeleton Key. J Am Coll Cardiol. 2015 Aug 4;66(5):561-77. doi: 10.1016/j.jacc.2015.05.066. PMID 26227196
- [Background] Menon V, Lincoln J. The Genetic Regulation of Aortic Valve Development and Calcific Disease. Front Cardiovasc Med. 2018 Nov 6;5:162. doi: 10.3389/fcvm.2018.00162. eCollection 2018. PMID 30460247
- [Background] Kostyunin AE, Yuzhalin AE, Ovcharenko EA, Kutikhin AG. Development of calcific aortic valve disease: Do we know enough for new clinical trials? J Mol Cell Cardiol. 2019 Jul;132:189-209. doi: 10.1016/j.yjmcc.2019.05.016. Epub 2019 May 25. PMID 31136747
- [Background] Small A, Kiss D, Giri J, Anwaruddin S, Siddiqi H, Guerraty M, Chirinos JA, Ferrari G, Rader DJ. Biomarkers of Calcific Aortic Valve Disease. Arterioscler Thromb Vasc Biol. 2017 Apr;37(4):623-632. doi: 10.1161/ATVBAHA.116.308615. Epub 2017 Feb 2. PMID 28153876
- [Background] Chin CW, Pawade TA, Newby DE, Dweck MR. Risk Stratification in Patients With Aortic Stenosis Using Novel Imaging Approaches. Circ Cardiovasc Imaging. 2015 Aug;8(8):e003421. doi: 10.1161/CIRCIMAGING.115.003421. No abstract available. PMID 26198161
- [Background] Aggarwal SR, Clavel MA, Messika-Zeitoun D, Cueff C, Malouf J, Araoz PA, Mankad R, Michelena H, Vahanian A, Enriquez-Sarano M. Sex differences in aortic valve calcification measured by multidetector computed tomography in aortic stenosis. Circ Cardiovasc Imaging. 2013 Jan 1;6(1):40-7. doi: 10.1161/CIRCIMAGING.112.980052. Epub 2012 Dec 10. PMID 23233744
- [Background] Clavel MA, Messika-Zeitoun D, Pibarot P, Aggarwal SR, Malouf J, Araoz PA, Michelena HI, Cueff C, Larose E, Capoulade R, Vahanian A, Enriquez-Sarano M. The complex nature of discordant severe calcified aortic valve disease grading: new insights from combined Doppler echocardiographic and computed tomographic study. J Am Coll Cardiol. 2013 Dec 17;62(24):2329-38. doi: 10.1016/j.jacc.2013.08.1621. Epub 2013 Sep 24. PMID 24076528
- [Background] Pawade T, Clavel MA, Tribouilloy C, Dreyfus J, Mathieu T, Tastet L, Renard C, Gun M, Jenkins WSA, Macron L, Sechrist JW, Lacomis JM, Nguyen V, Galian Gay L, Cuellar Calabria H, Ntalas I, Cartlidge TRG, Prendergast B, Rajani R, Evangelista A, Cavalcante JL, Newby DE, Pibarot P, Messika Zeitoun D, Dweck MR. Computed Tomography Aortic Valve Calcium Scoring in Patients With Aortic Stenosis. Circ Cardiovasc Imaging. 2018 Mar;11(3):e007146. doi: 10.1161/CIRCIMAGING.117.007146. PMID 29555836
- [Background] Glasziou P, Irwig L, Deeks JJ. When should a new test become the current reference standard? Ann Intern Med. 2008 Dec 2;149(11):816-22. doi: 10.7326/0003-4819-149-11-200812020-00009. PMID 19047029
- [Background] Messika-Zeitoun D, Aubry MC, Detaint D, Bielak LF, Peyser PA, Sheedy PF, Turner ST, Breen JF, Scott C, Tajik AJ, Enriquez-Sarano M. Evaluation and clinical implications of aortic valve calcification measured by electron-beam computed tomography. Circulation. 2004 Jul 20;110(3):356-62. doi: 10.1161/01.CIR.0000135469.82545.D0. Epub 2004 Jul 12. PMID 15249504
- [Background] Baumgartner H, Falk V, Bax JJ, De Bonis M, Hamm C, Holm PJ, Iung B, Lancellotti P, Lansac E, Rodriguez Munoz D, Rosenhek R, Sjogren J, Tornos Mas P, Vahanian A, Walther T, Wendler O, Windecker S, Zamorano JL; ESC Scientific Document Group. 2017 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2017 Sep 21;38(36):2739-2791. doi: 10.1093/eurheartj/ehx391. No abstract available. PMID 28886619
- [Background] Ajlan M, Ahmed A, Alskaini AM, Abukhaled NF, Alsaileek A, Ajlan A, Sulaiman IF, Al-Mallah MH. The reproducibility of coronary artery calcium scoring on different software platforms. Int J Cardiol. 2015;187:155-6. doi: 10.1016/j.ijcard.2015.03.133. Epub 2015 Mar 19. No abstract available. PMID 25828343
- [Background] Weininger M, Ritz KS, Schoepf UJ, Flohr TG, Vliegenthart R, Costello P, Hahn D, Beissert M. Interplatform reproducibility of CT coronary calcium scoring software. Radiology. 2012 Oct;265(1):70-7. doi: 10.1148/radiol.12112532. Epub 2012 Jul 6. PMID 22771886
- [Background] Baumgartner H Chair, Hung J Co-Chair, Bermejo J, Chambers JB, Edvardsen T, Goldstein S, Lancellotti P, LeFevre M, Miller F Jr, Otto CM. Recommendations on the echocardiographic assessment of aortic valve stenosis: a focused update from the European Association of Cardiovascular Imaging and the American Society of Echocardiography. Eur Heart J Cardiovasc Imaging. 2017 Mar 1;18(3):254-275. doi: 10.1093/ehjci/jew335. PMID 28363204